CLINICAL TRIAL: NCT05703360
Title: Effectiveness of Audiovisual Stimulation in Immersive Virtual Reality to Improve Visual Perception and Driving Performance: a Pilot Study
Brief Title: Effectiveness of AV-stimulation in Immersive VR to Improve Visual Perception and Driving Performance
Acronym: Re:DriVR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 22-5914
Record Dates: First submitted 2023-01-13; First posted 2023-01-30 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Stroke; Visual Impairment; Low Vision; Virtual Reality; Visual Spatial Processing; Visual Field Defect; Visual Processing Speed; Cognitive Impairment; Driving Impaired
MeSH Terms: conditions — Stroke; Vision Disorders; Vision, Low; Spatial Processing; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Interventional, pragmatic, cross-over, single-blind, multi-centre study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Waitlist Group (Experimental): Those randomly assigned to the waitlist group will complete initial inclusion tests and baseline tests at Visit 1. They will receive no intervention during Period 1 (week 1-6) and then repeat baseline tests at Visit 2. Next they will perform the VR audiovisual stimulation during Period 2 (week 7-12) and then repeat baseline tests post-intervention at Visit 3.
  Interventions: Device: Audiovisual Stimulation
- VR Intervention First (Experimental): Those randomly assigned to the intervention-first group will complete initial inclusion tests and baseline tests at Visit 1. They will perform the VR audiovisual stimulation during Period 1 (week 1-6) and then repeat baseline tests at Visit 2. They will receive no intervention during Period 2 (week 7-12) and then repeat baseline tests at Visit 3.
  Interventions: Device: Audiovisual Stimulation

INTERVENTIONS:
Device: Audiovisual Stimulation — The device application involves the 3D multiple-object-tracking (3D-MOT) paradigm composed of 8 high-contrast spheres which are adapted to the visual ability of participant (luminosity and size). The initial speed of the spheres is adjustable and determined during the inclusion visit.
  One or more of the spheres is temporarily highlighted (target). Then all 8 spheres move for 20 seconds following random linear paths, bouncing on one another and on the walls of a virtual 3D cube when collisions occur. After 20 seconds, the movement stops and the participant is asked to select, using the hand controller, the initially highlighted target(s) among the 8 spheres. If the selection is correct the speed of the spheres in the next trial is increased. If the selection is incorrect the speed of the spheres in the next trial is decreased.
  Based on performance, stimulations will be adjusted to change difficulty level (e.g. changing backgrounds, number of cued balls, etc.)

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of an immersive virtual-reality (IVR) based stimulation program, in improving visual perception for people who have lost their driver's license due to perceptual or cognitive impairments.

The main questions it aims to answer are:

1. Can the 6-week IVR stimulation program help improve driving performance?
2. Will participants experience improvement in visual detection and perception after training?

Study Design Summary:

* Participants will be randomized into a waitlist group or intervention-first group
* The VR-based intervention will consist of training every 2 days for six weeks
* Waitlist group will wait 6 weeks before starting intervention at study midpoint (week 7)
* Intervention-first group will begin with intervention (week 1-6) and then stop intervention at study midpoint
* Participants will complete tests related to driving performance, visual attention, and visual fields at the start of study, midpoint, and end of study

Researchers will analyze data for changes from baseline in outcome measures.

DETAILED DESCRIPTION:
This clinical trial will be an interventional, cross-over, single blind, randomized, supportive care, single-center study lasting 12 weeks with a target recruitment of 30 participants.

SCREENING AND BASELINE TESTS

Potential participants will be identified from patients receiving routine care at Toronto Western Hospital by their ophthalmologist. After obtaining informed consent and screened for inclusion, the research coordinator will set up appointments for each participant to complete baseline tests related to driving performance, visual attention, and visual fields. Participants will also practice the IVR program and be assessed for IVR sensitivity, or cybersickness, using the Virtual-Reality Induced Symptoms and Effects (VRISE) questionnaire.

Participants will be randomized into a Waitlist group or Intervention-First group. The Intervention-First group will be given a head-mounted display (HMD) to take home for training.

INTERVENTION (Week 1 - 12)

Period 1 (Week 1-6):

* Waitlist Group has no intervention
* Intervention-First group trains at home every 2 days using HMD

All participants are booked for their second appointments to repeat baseline tests once Period 1 is complete. Intervention-first group will return their HMD to the researchers and Waitlist group will be given their HMD to take home.

Period 2 (Week 7-12)

* Waitlist Group trains at home every 2 days using HMD
* Intervention-First group has no intervention

All participants are booked for their third appointments to repeat baseline tests once Period 2 is complete. Waitlist group will return their HMD to researchers.

POST-INTERVENTION

Analysis of outcome measures:

1. Period 1 (Waitlist Group vs Intervention-First Group)
2. Waitlist Group (Period 1 vs Period 2)
3. Intervention-First Group (Period 1 vs Period 2)

ELIGIBILITY:
Inclusion Criteria:

* Male and female > 25 years old.
* Visual field defects due to TBI or stroke
* BCVA ≥ 20/50.
* Previously held a valid driving license and were active drivers.
* Ability to follow the visual and auditory stimuli and training instructions.
* Online auditory test positive (-5dBHL to 60dBHL range) at 125 Hz (for research purposes only)
* Home Wi-Fi access.

Exclusion Criteria:

* Both eyes with media opacity that impairs visual field testing.
* Inability to perform during testing and training.
* Cognitive/motor condition incompatible with driving simulator and/or VR.
* Recreational or medicinal consumption of psychoactive drugs.
* 3 consecutive VRISE scores < 25 at inclusion.
* History of vertigo or dizziness.
* Visual neglect.
* Prior/current vision rehabilitation interventions.
* Photosensitive epilepsy.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in braking response (sec) | Initial visit (day 0), End of Period 1 (day 43), End of Period 2 (day 86)
  Driving performance will be assessed at the DriverLab, a driving simulator located at KITE-UHN under the supervision of the research team members.
Changes from baseline in collisions (total #) | Initial visit (day 0), End of Period 1 (day 43), End of Period 2 (day 86)
  Driving performance will be assessed at the DriverLab, a driving simulator located at KITE-UHN under the supervision of the research team members.
Changes from baseline in lane keeping (meters of deviations/departures) | Initial visit (day 0), End of Period 1 (day 43), End of Period 2 (day 86)
  Driving performance will be assessed at the DriverLab, a driving simulator located at KITE-UHN under the supervision of the research team members.
Changes from baseline in speed variability (km/h) | Initial visit (day 0), End of Period 1 (day 43), End of Period 2 (day 86)
  Driving performance will be assessed at the DriverLab, a driving simulator located at KITE-UHN under the supervision of the research team members.
Changes from baseline in road rule violations (# and type) | Initial visit (day 0), End of Period 1 (day 43), End of Period 2 (day 86)
  Driving performance will be assessed at the DriverLab, a driving simulator located at KITE-UHN under the supervision of the research team members.

SECONDARY OUTCOMES:
Changes from baseline in visual attention and speed using Re:ViewD | Initial visit (day 0), End of Period 1 (day 43), End of Period 2 (day 86)
  This vision test will be completed within the VR headset and will measure visual processing speed, sustained visual attention, and divided visual attention. This is a VR version of the Useful Field of View (UFoV) test which has been extensively used to measure visual attention in healthy individuals and older adults with low vision.
  Outcome measures are time of display (ms) for 75% of correct responses.
Changes from baseline in visual fields | Initial visit (day 0), End of Period 1 (day 43), End of Period 2 (day 86)
  Visual fields are evaluated with the automated Humphrey Field Analysis III using Esterman binocular field test procedure at Toronto Western Hospital.
  Outcome measures are number of points seen among 120 points.
Simulator Sickness Questionnaire (SSQ) | Initial visit (day 0), End of Period 1 (day 43), End of Period 2 (day 86)
  The SSQ will be administered after each driving session to capture any feelings related to simulator sickness.
  The SSQ is a validated 16-item questionnaire that assesses various symptom categories of simulator sickness. Responses are made on a 4-point scale ranging from "not at all" (total score = 0) to "severe" (total score =235.62). A total score (TS) ≥ 150 corresponds to mild to severe symptoms. Three subscales within the SSQ specifically targeting feelings of nausea (SSQ-N), oculomotor disturbances (SSQ-O), and disorientation (SSQ-D) as well as a total score (SSQ-TS) can be calculated based on pre-defined factor weightings.
Virtual-Reality Induced Symptoms and Effects (VRISE) - initial screening | Initial visit (day 0)
  This questionnaire is made up of five (5) questions related to possible cybersickness symptoms and will be completed within the VR headset by using the hand controller. Participants will complete the VRISE immediately after being trained on how to use the VR intervention at the initial visit. The VRISE score ranges from 5 (very intense level of symptoms and effects) to 35 (very low level of symptom and effects).
Virtual-Reality Induced Symptoms and Effects (VRISE) - intervention period | Every other day with training session (Weeks 1-6 for Intervention-First Group, Weeks 7-12 for Waitlist Group)
  This questionnaire is made up of five (5) questions related to possible cybersickness symptoms and will be completed within the VR headset by using the hand controller. Participants will complete the VRISE immediately after being trained on how to use the VR intervention at the initial visit. The VRISE score ranges from 5 (very intense level of symptoms and effects) to 35 (very low level of symptom and effects).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Reber, PhD, Principal Investigator — University Health Network, Toronto; Lora Appel, PhD, Principal Investigator — York University; Jennifer Campos, PhD, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - KITE Research Institute, UHN, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario

REFERENCES:
- [Background] Saredakis D, Szpak A, Birckhead B, Keage HAD, Rizzo A, Loetscher T. Factors Associated With Virtual Reality Sickness in Head-Mounted Displays: A Systematic Review and Meta-Analysis. Front Hum Neurosci. 2020 Mar 31;14:96. doi: 10.3389/fnhum.2020.00096. eCollection 2020. PMID 32300295
- [Background] Richards E, Bennett PJ, Sekuler AB. Age related differences in learning with the useful field of view. Vision Res. 2006 Nov;46(25):4217-31. doi: 10.1016/j.visres.2006.08.011. Epub 2006 Oct 5. PMID 17027061